CLINICAL TRIAL: NCT00229372
Title: Prolonged Exposure Versus Treatment as Usual in Chronic Posttraumatic Stress Disorder Combat and Terror Related Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Prof. Joseph Zohar, Chaim Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SHEBA-02-2732-JZ-CTIL
Record Dates: First submitted 2005-09-28; First posted 2005-09-29 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics

INTERVENTIONS:
Behavioral: Prolonged Exposure (PE) therapy

SUMMARY:
Assessing the efficacy of Posttraumatic Stress Disorder (PE) treatment for chronic Posttraumatic Stress Disorder (PTSD)

ELIGIBILITY:
Inclusion Criteria:

* PTSD

Exclusion Criteria:

* Psychotic symptoms
* Dissociation
* Drug or Alcohol dependence

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nitza Nacasch, MD, Study Chair — Tel Aviv University; Joseph Zohar, MD, Principal Investigator — Tel Aviv University
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Derived] Nacasch N, Foa EB, Huppert JD, Tzur D, Fostick L, Dinstein Y, Polliack M, Zohar J. Prolonged exposure therapy for combat- and terror-related posttraumatic stress disorder: a randomized control comparison with treatment as usual. J Clin Psychiatry. 2011 Sep;72(9):1174-80. doi: 10.4088/JCP.09m05682blu. Epub 2010 Nov 16. PMID 21208581